CLINICAL TRIAL: NCT07241416
Title: A Multicenter, Randomized, Open-Label, Positive-Controlled Phase III Study of Rezvilutamide Combined With Androgen Deprivation Therapy (ADT) Versus Enzalutamide Combined With ADT for Treating Low-volume Metastatic Hormone Sensitive Prostate Cancer (mHSPC)
Brief Title: A Phase III Clinical Study of Rezvilutamide in Patients With Metastatic Hormone-Sensitive Prostate Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-PCa-III-021
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Hormone-sensitive Prostate Cancer (mHSPC)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rezvilutamide Tablets Group (Experimental)
  Interventions: Drug: Rezvilutamide Tablets
- Enzalutamide Soft Capsules Group (Active Comparator)
  Interventions: Drug: Enzalutamide Soft Capsules

INTERVENTIONS:
Drug: Rezvilutamide Tablets — Rezvilutamide tablets, oral administration.
  Arms: Rezvilutamide Tablets Group
Drug: Enzalutamide Soft Capsules — Enzalutamide soft capsules, oral administration.
  Arms: Enzalutamide Soft Capsules Group

SUMMARY:
This study aims to compare the efficacy and safety of rezvilutamide with enzalutamide in the treatment of patients with low-volume metastatic hormone sensitive prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participates in this clinical trial, with an understanding of the study procedures and signed informed consent;
2. Age ≥ 18 years;
3. Histologically or cytologically confirmed prostate adenocarcinoma without evidence of neuroendocrine differentiation or small cell features;
4. Metastatic hormone sensitive prostate cancer;
5. ECOG PS: 0-1;
6. Planned to receive and maintain ADT during the study period;
7. Adequate hepatic, renal, heart, and hematological functions;
8. Determined by the investigator to be able to comply with the study protocol;
9. Fertile subjects must use effective contraception or abstain from sexual activity and sperm donation until 3 months after last exposure to rezvilutamide or enzalutamide. Subjects must use condoms plus an additional effective contraceptive method during sexual activity with a fertile female partner throughout treatment and for 3 months post-treatment.

Exclusion Criteria:

1. Prior treatment with ADT, chemotherapy, surgery, external-beam radiotherapy, brachytherapy, radiopharmaceuticals, or investigational local therapy for metastatic prostate cancer, except as specifically allowed by the protocol;
2. Previous use of second-generation androgen receptor antagonists, ketoconazole, abiraterone acetate, or other investigational drugs inhibiting androgen synthesis for prostate cancer treatment; or plans to use any second-generation androgen receptor antagonist other than the study drug during the study treatment period;
3. Total PSA has decreased to undetectable levels at baseline;
4. Have participated in an interventional clinical trial or been treated with the following drugs in the past 4 weeks before randomization: 5-alpha reductase inhibitors, estrogen, progestin, and herbal products known to decrease PSA levels;
5. Planned to initiate any other anti-tumor therapies during the study;
6. Known history of hypersensitivity to rezvilutamide, enzalutamide, or any of their components;
7. Unable to swallow, chronic diarrhea or intestinal obstruction, or the presence of a variety of other factors that affect drug use and absorption;
8. History of seizure or certain conditions that may predispose to seizure;
9. Presence of clinically significant cardiovascular diseases within 6 months prior to randomization;
10. Any other malignancy within 5 years prior to randomization (except as specifically allowed by the protocol);
11. Active HBV or HCV infection;
12. History of immunodeficiency (including HIV-positive status, other acquired or congenital immunodeficiency disorders) or organ transplantation;
13. Any concomitant condition that, in the opinion of the investigator, would seriously jeopardize patient safety, confound study findings, or compromise the patient's ability to complete the study (e.g., hypertension inadequately controlled despite medication, severe diabetes, neurologic or psychiatric disorders, etc.) or any other circumstance.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Prostate Specific Antigen (PSA) undetectable rate based on central laboratory. | 6 months after randomization.
  Defined as the proportion of subjects with a total PSA level below 0.2 ng/mL in central laboratory testing within 6 months after randomization.

SECONDARY OUTCOMES:
PSA response rate based on local laboratory. | Up to approximately 5 years.
  Defined as the proportion of subjects who achieved a ≥50% or ≥90% reduction in PSA levels from baseline among those who had not initiated ADT treatment prior to randomization.
PSA undetectable rate based on local laboratory. | 6 months after randomization.
  Defined as the proportion of subjects with a total PSA level below 0.2 ng/mL in local laboratory within 6 months after randomization.
Objective response rate (ORR). | Up to approximately 5 years.
  The percentage of subjects with measureable disease at baseline who achieved a complete or partial response in their soft tissue disease using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria and PCWG3.
Radiographic progression-free survival (rPFS). | Up to approximately 5 years.
  Time from randomisation to radiologically confirmed progressive disease or death due to any cause.
Time to PSA progression based on local laboratory. | Up to approximately 5 years.
  Time from randomisation to the first time of PSA progression according to the criterion of PCGW3.
Time to castration-resistant prostate cancer (CRPC). | Up to approximately 5 years.
  Defined as the time from randomization to the first occurrence of castration-resistant event.
Overall survival (OS). | Up to approximately 5 years.
  Defined as the time from randomization to death due to any cause.
Adverse events (AEs). | Up to approximately 5 years.
  An AE is any untoward medical occurrence in a participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Medical Center of the Chinese People's Liberation Army (PLA) General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided